CLINICAL TRIAL: NCT01663558
Title: Anal Dysplasia Study of Men Who Have Sex With Men Living With HIV
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: funding not available
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23592103
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Anal Dysplasia; Human Papilloma Virus; HIV
Keywords: anal dysplasia; HPV; HIV; MSM
MeSH Terms: interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- imiquimod (Active Comparator): i. Each subject will use an imiquimod anal suppository three times weekly (overnight on Monday, Wednesday, Friday) for 12 weeks.
  ii. Each subject will be asked to abstain from receptive anal sex during therapy period (12 weeks).
  iii. If local imiquimod adverse effects are severe, a 7-day period off of treatment will be permitted.
  iv. During 12 week therapy period, each subject will be evaluated 2, 4, 8, and 12 weeks after starting therapy. At each visit, subject will complete a therapy questionnaire and undergo anal Pap, HRA with biopsies as indicated, and anal HPV testing.
  v. After therapy completed (12 weeks), subject will enter 12 month observation period.
  Interventions: Drug: imiquimod
- ablative (Active Comparator): i. Subject will be referred to colorectal surgeon, will complete a therapy questionnaire, and will be treated in accordance with treatment algorithm which is already in use.
  ii. Subject will be asked to abstain from receptive anal sex for 12 weeks after ablative therapy.
  iii. After therapy, subject will enter 12 month observation period.
  Interventions: Procedure: ablative
- Observation (No Intervention): i. Given lack of accepted guidelines and outcome data on dysplasia management, the study PI will thoroughly discuss risks and benefits of observation/monitoring and treatment of dysplasia.
  ii. If treatment is chosen, subject will be randomized to 1) ablative group, or 2) imiquimod group and begin therapy. Observation subjects will continue observation visits (observation questionnaire, anal Pap, HRA with biopsies as indicated, and anal HPV testing) every 3 months for 12 months (4 additional study visits).

INTERVENTIONS:
Drug: imiquimod
  Other Names: Aldara
  Arms: imiquimod
Procedure: ablative
  Arms: ablative

SUMMARY:
Context:

Men who have sex with men (MSM) are at increased risk for HPV-related anal neoplasia and anal squamous cell carcinoma; concomitant HIV infection roughly doubles that risk.

Objectives:

1. To compare the efficacy of ablative therapy to topical imiquimod therapy in the management of anal dysplasia in HIV-infected men.
2. To describe relationship between cytologic grade of anal dysplasia (as reported on screening anal Pap test) and pathologic grade reported on anal mucosa histopathologic examination.
3. To describe demographic, sexual practices, HPV-specific, and HIV-specific correlates of anal dysplasia.
4. To describe adverse effects associated with ablative therapy and topical imiquimod therapy.

Design:

Prospective, randomized controlled clinical trial. This will be a pilot study. All subjects will undergo baseline anal Pap, HRA with biopsies as indicated, and anal HPV testing. If AIN 2 or 3 is discovered on histopathologic examination, subject will be offered observation only or treatment. If he chooses treatment, he will be randomized to: 1) imiquimod anal suppositories three times weekly for 3 months, or 2) appropriate ablative therapy as determined by colorectal surgeon. During imiquimod treatment (not applicable to ablative group as their treatment will be completed in one visit) subjects will be followed for 2 weeks, 4 weeks, 8 weeks, and 12 weeks with anal Pap, HRA with biopsies as indicated, and anal HPV testing. After therapy completed in each treatment group, subjects will be followed for 1 month, 3 months, 6 months, 9 months, and 12 months post-therapy with anal Pap, HRA with biopsies as indicated, and anal HPV testing. Observation only subjects will be evaluated every 3 months with anal Pap, HRA with biopsies as indicated, and anal HPV testing for 12 months. We have chosen a goal of 30 subjects in each treatment group and 10 subjects in the observation only group based on the likelihood of enrolling a study of this type in a reasonable amount of time.

Main Outcome Measures:

1. Anal Pap cytologic grade, including regression and recurrence during course of study
2. HPV type in anal canal, including regression and recurrence during course of study
3. Anal histology, including regression and recurrence during course of study
4. Adverse effects experienced during treatment, recorded in symptom log

ELIGIBILITY:
Inclusion Criteria:

* Male gender, ≥18 years of age
* HIV-infected and taking ARVs with suppressed HIV VL (<48 copies/mL) on 2 consecutive measurements within the previous 6 months
* Any CD4 count will be considered appropriate for study
* Plasma INR < 1.5
* Plasma partial thromboplastin time (PTT) < 35s
* Blood WBC > 2.0x103/mm3 and absolute neutrophils count > 500
* Blood hemoglobin > 10.0 g/dL
* Blood platelet count > 50x103/mm3
* Serum total bilirubin < 6.0 mg/dL (subjects taking atazanavir-based ARV regimens may have elevated total bilirubin but are generally < 6)
* Blood aspartate aminotransferase (AST) < 100 U/L (<2 ULN)
* Blood alanine aminotransferase (ALT) < 130 U/L (<2 ULN)
* Serum creatinine < 1.5 mg/dL
* ECOG performance status < 3
* Tricare beneficiary

Exclusion Criteria:

* History of AIN
* Anal canal condyloma requiring surgical treatment
* Anal cancer (current or history of)
* History of prior anal surgery, including hyfrecation, excision, cryotherapy, photocoagulation
* Use of anticoagulants (warfarin, heparin, Pradaxa)
* Inability to attend study visits
* Participation in any other drug study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
cytologic grade | 3 months
  Anal Pap cytologic grade, including regression and recurrence during course of study

SECONDARY OUTCOMES:
HPV | 3 months
  HPV type in anal canal, including regression and recurrence during course of study

OTHER OUTCOMES:
histologic grade | 3 months
  Anal histology, including regression and recurrence during course of study

CONTACTS AND LOCATIONS:
Overall Officials: John D Malone, MD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- NMCSD, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No